CLINICAL TRIAL: NCT06785207
Title: Rethinking Rigidity: Development of a 3D-Printed Scoliosis Brace With Varying Flexibility
Acronym: 3DSCOLIBRACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Scoliosis Research Society (SRS) (Unknown)
Responsible Party: Principal Investigator, Megan Elizabeth Castille, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H-55196
Record Dates: First submitted 2025-01-16; First posted 2025-01-21 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Scoliosis Idiopathic Adolescent Treatment
Keywords: 3D-printed scoliosis brace; scoliosis brace; scoliosis bracing; 3D-printing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 3D-printed brace (Experimental): Enrolled participants will be fit with a 3D printed brace. The brace will be made using the exact same shape as their current brace. The fitting procedures will also remain the same.
  Interventions: Device: 3D-printed scoliosis brace

INTERVENTIONS:
Device: 3D-printed scoliosis brace — Scoliosis brace will be 3D printed using a Filament Innovations Icarus printer and the material CPX. There will be corrugations where extra strength is needed. The brace will be made using the same shape as the participant's current brace to minimize variables at play.
  According to Sec. 890.3490 of the Code of Federal Regulations Title 21, scoliosis braces are Class I devices, requiring only general controls. This device is exempt from the premarket notification procedures in subpart E of part 807 of this chapter, subject to the limitations in § 890.9. The device is also exempt from the current good manufacturing practice requirements of the quality system regulation in part 820 of this chapter, with the exception of § 820.180, regarding general requirements concerning records and § 820.198, regarding complaint files.

SUMMARY:
Scoliosis bracing is an effective treatment method for idiopathic scoliosis, but only if worn consistently for many hours a day. Unsurprisingly, brace discomfort is a significant deterrent against treatment adherence. For decades, custom braces for idiopathic scoliosis have been fabricated using one of three materials - copolymer, polypropylene, or polyethylene. The application of the biomechanical principles behind bracing have improved over the years, but the materials have not. The investigators' goal is to expand fabrication options by testing a 3D-printed scoliosis brace with variable flexibility. The aim is to improve patients' perceived brace comfort.

After optimizing the brace design, the investigators will collect patient feedback about the design from currently braced participants. These participants understand what a standard brace feels like and will provide impactful feedback.

DETAILED DESCRIPTION:
After optimizing the brace design, the investigators will collect patient feedback about the design from currently braced participants. Once a participant enrolls in the study, the 3D printed brace will be made using the exact same shape as their current brace. The standard fabrication process includes the following:

1. Certified orthotist completes a full evaluation
2. Taking a scan of the patient's body
3. Modifying, or editing, the patient's body shape using Computer-Aided-Design and applying corrective pressures against the apex of the scoliotic curve
4. Carving a positive foam model of the modified shape and thermoforming the polypropylene plastic over the positive foam model

These steps were already completed to make the participant's current brace, which has been deemed acceptable by their medical team, including the PI and Dr. Timothy Borden. To reduce the number of variables present, the 3D printed brace will be made using the exact same shape as their current brace. The only difference is the fabrication technique (step 4). Instead of carving a foam mode and thermoforming, the exact brace shape will be directly 3D printed. Therefore, no additional x-rays, scans, or measurements are required from the participants. The standard fabrication process and research activities are outlined in attachment titled "Fabrication Process Outline."

Once the 3D printed brace has been fabricated, the participant will come in to be fit with the brace. A standard fitting involves trimming the brace, adding straps, heating and flaring to improve comfort, and potentially adding padding. The PI is a scoliosis bracing specialist and will be the lead orthotist during the fitting process to ensure that best practices are followed.

Following the fitting, the participant will provide test out the 3D printed brace for comfort by performing a series of tasks. The activities will include the following: sitting in a chair, picking an item up from the floor while standing, picking an item up from the floor while sitting, stepping onto a stool, jogging in place for 10s, performing the hula hoop Wii-fit game, lying down on an exam table, and donning shoes. All data collection will take place via the survey platform Qualtrics.

If the participants feel comfortable in the brace and pass a skin check, the participants will then take the brace home and wear it for 1 week. They will return for the 1-week follow-up appointment and complete the study at this time. They will provide feedback about the 3D printed brace through a semi-structured interview (recorded using BCM Zoom Platform) and complete a survey (Qualtrics). They will return the brace, marking the end of the study.

Total duration of study participation ranges from 2 weeks - 6 weeks. The time commitment required from the participant is no more than 8 hours. The timelines are outlined below:

1. Participant enrollment during appointment at Align Clinic (complete consent forms, demographic survey, baseline testing). Study-related activities will take approximately 30-60 minutes
2. 3D printed brace fabrication. Nothing required of participants. Fabrication will take roughly 1-4 weeks
3. Brace fitting. Participant will come to the office to be fit with the 3D-printed brace. Fitting will take roughly 1-4 hours
4. Activity series in 3D printed brace. Will occur on the same day as the fitting. Testing will take approximately 30 minutes
5. Follow-up appointment one week after the fitting. 3D printed brace is returned, marking the end of the study. Study activities (semi-structured interview, survey) will take 30-60 minutes.

Standard of care will be maintained throughout the study. The only activities outside of the standard of care are the semi-structured interview, study surveys, and performance of tasks. While the goal of the study is to elevate the 3D printed materials, the investigators will still be following the standard of care for 3D printing.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of juvenile idiopathic scoliosis or adolescent idiopathic scoliosis
2. Have a Cobb angle between 20-40 degrees
3. Are between ages 8-18
4. Present as Risser 2+ on x-ray
5. Currently wear a traditionally fabricated scoliosis brace
6. Have good brace adherence in current brace (self-reported to be 75% of prescribed time)
7. Be an established patient of Align Clinic and Dr. Timothy Borden
8. Speak English (survey and semi-structured interview will only be available in English)
9. Assent and receive parental consent

Exclusion Criteria:

1. Have a diagnosis other than juvenile idiopathic scoliosis or adolescent idiopathic scoliosis
2. Have a Cobb angle outside the range of 20-40 degrees
3. Present as Risser 0 or 1
4. Do not currently wear a traditionally fabricated scoliosis brace
5. Have poor adherence in their current brace
6. Do not speak English
7. Are not willing participate in the study

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceived brace comfort | Comparing baseline comfort measures at enrollment (current brace) to comfort measures in 3D-printed brace at fitting (roughly 4 weeks after enrollment)
  Participants will complete a series of tasks (sitting down, putting shoes on, stepping onto stool, etc.) in their current brace and in the 3D-printed scoliosis brace. Each task will be completed three times and researchers will be blinded to participant responses. A Wilcoxon signed-rank test will compare 3D printed brace comfort to baseline measures.

SECONDARY OUTCOMES:
Semi-structured interview | Conducted at one-week follow-up appointment
  A semi-structured interview will be performed to understand the differences between the two braces. Systematic coding procedures (e.g., open, axial, and selective coding) will be conducted by the research team.

OTHER OUTCOMES:
Survey about perceived brace fit and comfort | Completed at one-week follow-up appointment
  Participants will answer a survey about their experience during the one-week trial with the 3D-printed brace. The survey will ask about comfort, preferences, design, etc.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Align Clinic, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nathan P, Chou SM, Liu G. A review on different methods of scoliosis brace fabrication. Prosthet Orthot Int. 2023 Aug 1;47(4):424-433. doi: 10.1097/PXR.0000000000000195. Epub 2023 Jan 31. PMID 36723398
- [Background] Ronca A, Abbate V, Redaelli DF, Storm FA, Cesaro G, De Capitani C, Sorrentino A, Colombo G, Fraschini P, Ambrosio L. A Comparative Study for Material Selection in 3D Printing of Scoliosis Back Brace. Materials (Basel). 2022 Aug 19;15(16):5724. doi: 10.3390/ma15165724. PMID 36013868